CLINICAL TRIAL: NCT06547177
Title: The Effect of Nutrition and Fluid Intake in the First Stage of Labor on Maternal and Fetal Outcomes
Brief Title: The Effect of Nutrition and Fluid Intake in the First Stage of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hilal Yuvacı (Other)
Responsible Party: Sponsor-Investigator, Hilal Yuvacı, Assoc. Prof. Dr., Sakarya University
Organization: Sakarya University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: fluid intake in labor
Record Dates: First submitted 2022-12-20; First posted 2024-08-09 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Labor Pain; Nutrient Intake; Fluid Therapy
Keywords: Labor; nutrition; fluid; labor pain; maternal outcome; fetal outcome
MeSH Terms: conditions — Labor Pain | interventions — Fruit and Vegetable Juices; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (No Intervention): Pregnant women in the study's control group will not be subjected to any application other than routine hospital practices. They will not consume oral liquid or solid food, and their fluid needs will be met with 125 ml/hour of intravenous(iv) fluid (5% dextrose).
- Fruit juice and water group (Experimental): Fruit juice (100 ml juice once in the first hour of admission to the delivery room during the latent phase) = (cherry/apple juice, 100 ml, 50-54 kcal), then every 4 hours. It will be given in 100 ml. In addition, they will be allowed to take small amounts of water. (Total fluid intake will be recorded)
  Interventions: Other: fruit juice
- Water group (Experimental): Water (as much as desired in 100 ml containers during the latent phase) (total water amount will be recorded). Pregnant women in all groups will not take oral fluids after transitioning to the active phase (> 6 cm cervical dilatation).
  Interventions: Other: fruit juice

INTERVENTIONS:
Other: fruit juice — During labor, one group will follow the routine while the water group will only take water and fruit juice group will take water and fruit juice.
  Other Names: water
  Arms: Fruit juice and water group; Water group

SUMMARY:
Birth is a process that requires large amounts of energy. As a result of skeletal and smooth muscle contractions at birth, the body's basal metabolic rate, energy requirement, hydration requirement, and insensible fluid loss are significantly increased. Information regarding the safety and effectiveness of increased hydration during labor is still controversial. There is no consensus on whether this hydration should be given with intravenous solutions or orally. The study aims to determine the effect of fluid intake in labor on the delivery process, maternal-fetal outcomes, and postpartum satisfaction of the mother.

DETAILED DESCRIPTION:
Method of Study: The study was planned as a randomized controlled experimental study to evaluate the effect of fluid intake during labor on mothers and babies.

Location and Characteristics of the Research: The research will be conducted in the delivery room of Sakarya Training and Research Hospital.

Population and Sample of the Study: The research will consist of pregnant women who apply to Sakarya Training and Research Hospital with signs of the onset of labor and will have an expected vaginal delivery in the delivery room. Annually, 7000-8000 women give birth in the hospital, and approximately 50% have an expected vaginal delivery. All pregnant women who met the sampling criteria and volunteered to participate in the study during the study's implementation will be included. The research will be carried out in 3 groups experimental and control groups. The study will be conducted with a total of 90 pregnant women, 30 of whom are in each group.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the research
* Agreeing to abide by the protocol
* Being able to read and write,
* Ages 18-35 years
* 37-40 Pregnancy weeks
* First pregnancy,
* Single fetus
* BMI ≤ 28,
* Head presentation
* Cervical dilatation of <6 cm or less (latent phase)
* Height ≥ 1.50 cm

Exclusion Criteria:

* Communication barriers (speech, hearing, mental),
* Disability (physical or mental problem, drug use),
* Chronic diseases (hypertension, diabetes, etc),
* Gastrointestinal problems before and during pregnancy
* Comply with the fluid intake protocol during labor,
* Pregnant women who are scheduled for elective cesarean section
* Pregnant women considered to be at immediate cesarean risks, such as diabetic pregnant women with cephalopelvic incompatibility, multiple pregnancies, preeclampsia, and macrosomic fetus

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Maternal outcome | The duration of the labor will measured from the latent phase of labor to birth.
  During the research, duration of the latent and active phase of labor will be recorded.
Maternal pain outcome | The study will be conducted from the latent phase of labor to birth.
  A visual analogue scale (VAS) was used to measure the levels of labor pain. VAS scores will be recorded from the latent phase of labor to birth.The VAS was a 0 to 100 mm line (from no pain to worst imaginable pain). Over 60 mm on the VAS indicates severe pain, moderate pain ranges from 40 - 60 mm and mild pain is under 40 mm. The higher scores implied the higher level of pain.
fetal outcomes | APGAR scores will be recorded after birth.
  The Apgar score is a standardized assessment of a neonate's status immediately after birth and the response to resuscitation efforts and remains the gold standard for evaluating neonates.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal Uslu Yuvacı, Principal Investigator — Sakarya University School of Medicine
Locations (1):
- Sakarya University School of Medicine, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT06547177/Prot_001.pdf